CLINICAL TRIAL: NCT06477835
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase 3 Study to Evaluate the Efficacy and Safety of SIM0718 in Adult and Adolescent Patients With Moderate to Severe Atopic Dermatitis
Brief Title: A Study to Evaluate the Efficacy and Safety of SIM0718 in Adult and Adolescent Patients With Moderate to Severe Atopic Dermatitis
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Simcere Pharmaceutical Co., Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SIM0718-302
Record Dates: First submitted 2024-06-14; First posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Active Comparator): During the placebo-controlled double-blind treatment phase, subjects were randomized 1:1 to the following treatment groups:
  • Test group: SIM0718 300 mg SC with loading dose of 600 mg on Day 1.
  During the W16-W52 Maintenance Period:
  • All subjects were dosed SC at 300 mg SIM0718.
  Interventions: Biological: SIM0718 Injection
- Control group (Placebo Comparator): During the placebo-controlled double-blind treatment phase, subjects were randomized 1:1 to the following treatment groups:
  • Volume-matched placebo SC, placebo loading dose on Day 1.
  During the W16-W52 Maintenance Period:
  • All subjects were dosed SC at 300 mg SIM0718.
  Interventions: Biological: SIM0718 Injection

INTERVENTIONS:
Biological: SIM0718 Injection — Subjects who meet entry criteria will be randomized in a 1:1 ratio to receive either SIM0718 or matching placebo,Q2W, SC until Week 16. At the Week 16 visit, subjects in the placebo group will be transferred to SIM0718 300 mg Q2W after completing safety and efficacy assessments. Subjects who were originally treated with 300 mg Q2W of SIM0718 will continue on their original treatment regimen.

SUMMARY:
This study will evaluate the efficacy and safety of SIM0718 in adolescents (12- < 18 years) and adults (18-75 years) with moderate to severe AD.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled multicenter clinical study to evaluate the efficacy and safety of SIM0718 in adolescents (12- < 18 years) and adults (18-75 years) with moderate to severe AD. Subjects who meet entry criteria will be randomized to receive either SIM0718 or matching placebo.The study includes a screening period, a treatment period and a follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 12 and ≤ 75 years, male or female, and body weight ≥ 40 kg at the screening visit.
2. Diagnosis of atopic dermatitis at screening (according to the American Academy of Dermatology Concordance Criteria, 2014), and: 1) Adult diagnosed AD for ≥ 12 months and adolescent diagnosed AD for ≥ 6 months prior to screening; 2) Inadequate response or intolerance to topical medications, or is medically inappropriate for topical treatment judged by the investigator within 6 months prior to Screening; 3) At Screening and Baseline,IGA score ≥3; 4)At Screening and Baseline, EASI score ≥ 16; 5) At Screening and Baseline,total AD involvement ≥ 10% BSA; 6) Baseline peak pruritus NRS score ≥ 4.

Exclusion Criteria:

1. Not enough washing-out period for previous therapy.
2. History of any of the following:

1) History of significant immune reactions (eg, serum sickness, anaphylaxis, or delayed hypersensitivity) to any other biologic agent or any excipient of SIM0718; 2) Presence of other active skin comorbidities other than AD that may interfere with study assessments, such as scabies, skin lymphoma, or psoriasis; 3) Active keratoconjunctivitis and atopic keratoconjunctivitis at screening; or previous history of recurrent keratoconjunctivitis and atopic keratoconjunctivitis; 4) Patients with active tuberculosis (TB), latent TB, or a history of nontuberculous mycobacterial infection at screening; 5) HBsAg positive at screening; or HBcAb positive with HBV-DNA positive; or hepatitis C antibody positive with HCV RNA polymerase chain reaction positive; or HIV serology positive; 6) Systemic treatment with antibiotics, antivirals, antiparasitic agents, antiprotozoal agents, or antifungal agents for infections within 4 weeks prior to baseline, or superficial skin infections within 1 week prior to baseline that could interfere with study assessments (subjects could be re-screened after resolution of infection); 7) History of parasitic infection within 6 months prior to baseline; 8) According to the investigator 's judgment, known or suspected history of immunosuppression within 6 months prior to baseline, including but not limited to history of invasive opportunistic infections, such as aspergillosis, coccidioidomycosis, histoplasmosis, HIV, listeriosis, pneumocystis disease or tuberculosis; or the presence of abnormal frequent recurrent or persistent infections; 9) History of malignancy within 5 years prior to screening.

3. Planned major surgical procedures during the study.

4. History of alcohol or drug abuse within 2 years before screening.

5. Any other condition that, in the judgment of the investigator, would make participation in this study inappropriate.

6. Female subjects of childbearing potential, who experience any of the following

* Positive serum pregnancy test or positive urine pregnancy test before baseline
* Pregnant or breastfeeding women, or women planning to become pregnant or breastfeeding during the study who are unwilling to use at least one highly effective form of birth control throughout the study and for 90 days after the last dose of study drug.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
EASI-75 at week 16 | Day1-Week16
  Proportion of subjects achieving EASI-75 at week 16.
IGA score at week 16 | Day1-Week16
  Proportion of subjects with IGA score of 0 or 1 and a reduction of IGA score by ≥2 points from baseline at week 16.

SECONDARY OUTCOMES:
EASI-75 at each visit | Day1-Week52
  Proportion of subjects achieving EASI-75 at each visit
EASI-50 at each visit | Day1-Week52
  Proportion of subjects achieving EASI-50 at each visit
EASI-90 at each visit | Day1-Week52
  Proportion of subjects achieving EASI-90 at each visit
NRS score | Day1-Week52
  Percent change of NRS score from baseline
BSA | Day1-Week52
  Body surface area (BSA) of involvement of atopic dermatitis
DLQI | Day1-Week52
  Changes from baseline in Dermatology Life Quality Index (DLQI)
Incidence of adverse events (AEs) | Day1-Week60
  Incidence of adverse events (AEs), abnormal physical examinations, abnormal vital signs, abnormal ECG, and abnormal lab testing

CONTACTS AND LOCATIONS:
Overall Officials: Jianzhong Zhang, Principal Investigator — Peking University People's Hospital; Cheng Zhou, Principal Investigator — Peking University People's Hospital

IPD SHARING:
Plan to Share IPD: No